CLINICAL TRIAL: NCT07127432
Title: The Effect of Storytelling Caterpillar Use on Pain, Anxiety, and Parental Satisfaction During Blood Draw in Children Aged 3 to 6 Years: A Randomized Controlled Trial
Brief Title: Storytelling Caterpillar - Pain, Anxiety, and Satisfaction
Acronym: SC-PAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Collaborators: Çam Sakura Şehir Hastanesi (Unknown)
Responsible Party: Principal Investigator, Eysan Hanzade Umac, Teaching Assistant, Koç University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KOCUNIV
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Children, Preschool; Pain and Anxiety
Keywords: distraction; satisfaction; storytelling; distraction techniques
MeSH Terms: conditions — Pain; Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Parallel assignment randomized controlled trial in which participants are allocated to either an intervention group receiving the Storytelling Caterpillar distraction tool during venous blood draw or a control group receiving standard care. Outcomes are compared between groups.
Masking Description: No masking was applied due to the nature of the intervention; both participants and outcome assessors were aware of group assignments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-Storytelling Caterpillar (Experimental): Children in the intervention group were introduced to the 'Storytelling Caterpillar' toy, a colorful, interactive device with music and narrated stories designed to provide visual, auditory, and tactile stimulation. The toy was activated one minute before the blood draw procedure, with the child seated on the parent's lap. The storytelling continued throughout the procedure to divert the child's attention and reduce pain and anxiety.
  Interventions: Device: The Storytelling Caterpillar
- Standard care group (No Intervention): Children in the control group received standard care during the blood draw procedure, which included parental presence and verbal reassurance provided by the nurse. No additional distraction or intervention was applied.

INTERVENTIONS:
Device: The Storytelling Caterpillar — The Storytelling Caterpillar is a plastic toy measuring 19.5 × 5.5 × 25.5 cm and is recommended for use in children aged 1-6 years. It is designed in the form of a storybook and includes interactive f
  Arms: Intervention-Storytelling Caterpillar

SUMMARY:
This randomized controlled trial aims to evaluate the effect of using the "Storytelling Caterpillar" toy on pain, anxiety, and parental satisfaction during blood draw procedures in children aged 3 to 6 years. The Storytelling Caterpillar is a colorful, interactive toy that combines visual, auditory, and tactile stimuli to engage children's attention through storytelling and music. The study will compare an intervention group, where the toy is used during the blood draw, with a control group receiving standard care without the toy. Outcomes will include pain levels assessed using the FLACC scale, anxiety levels evaluated with the Visual Analog Scale for Anxiety (VAS-A), and parental satisfaction measured using a VAS satisfaction score. The results are expected to provide evidence on the effectiveness of storytelling-based distraction in improving the procedural experience for children and their parents.

DETAILED DESCRIPTION:
Fear of medical procedures can reduce children's participation in healthcare, hinder access to medical services, and negatively impact the treatment process. Needle-related interventions such as blood draws, injections, and intravenous catheter insertions are often perceived by children as painful, frightening, and potentially traumatic. These experiences are more common in children with chronic illnesses, where the anticipation of pain often leads to heightened anxiety. Pediatric nurses, who frequently perform these invasive procedures, play a critical role in minimizing pain and anxiety during medical care. In addition to pharmacological methods, non-pharmacological approaches are commonly used due to their ease of application and absence of side effects. Among these, distraction techniques are widely preferred. These methods aim to divert the child's attention away from the procedure to a more engaging stimulus, thereby reducing pain, fear, and anxiety. Such interventions not only alleviate acute symptoms but also enhance treatment compliance and overall outcomes. Furthermore, distraction strategies can help reduce parental anxiety.

It is recommended that distraction tools used in pediatric settings incorporate both visual and auditory stimuli. One such method is storytelling with visual materials. Storytelling involves conveying narratives through words, sounds, and images, helping children process experiences and manage emotional responses by transforming events into coherent narratives. As a non-invasive, cost-effective, and easy-to-use technique, storytelling can reduce pain and anxiety in hospitalized children. Stories also serve as models for teaching values and coping strategies, providing insight at both conscious and subconscious levels. By focusing the child's attention on the story rather than the procedure, storytelling shifts perception away from the painful stimulus. Immersion in storytelling may also stimulate physiological responses that contribute to reduced pain and fear. Previous studies have shown that storytelling in pediatric populations can lead to lower anxiety and pain levels during medical procedures.

In light of this, the present study aimed to evaluate the effectiveness of a developmentally appropriate distraction tool-the Storytelling Caterpillar-in reducing pain and anxiety during blood draw procedures in children aged 3 to 6 years. This colorful, music-playing, interactive toy is designed to tell stories while stimulating the visual, auditory, and tactile senses, making it particularly engaging for this age group. It was expected that the use of the Storytelling Caterpillar would not only help reduce children's procedural anxiety and pain but also support pediatric nurses by facilitating the procedure and increasing the child's cooperation. Additionally, improvements in parental satisfaction were anticipated as a result of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* being between 3 and 6 years of age,
* having a parent who voluntarily agreed to participate in the study.

Exclusion Criteria:

* having a chronic illness requiring regular invasive procedures,
* having received analgesics within the past 2 hours,
* having experienced a seizure within the past 2 hours,
* using antiepileptic medication,
* having a body temperature above 37.5°C
* not having parental consent,
* being agitated at the time of the procedure,
* having any auditory or visual impairments.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Pain was measured once - immediately after the procedure (experienced pain).
  Pain was assessed using the Wong-Baker FACES Pain Rating Scale, a validated self-report tool for children. The scale consisted of six illustrated faces ranging from a happy face (score of 0, indicating "no pain") to a crying face (score of 10, indicating "worst pain"). Children were asked to choose the face that best represented the pain they felt during the procedure.
Fear | Fear was measured twice - immediately before the procedure (anticipated fear) and during the procedure (observed fear).
  The child's fear level was assessed using the Children's Fear Scale, a 5-face pictorial scale scored from 0 ("no fear") to 4 ("maximum fear").
Anxiety Level | Anxiety was measured twice - immediately before the procedure (anticipated anxiety) and immediately after the procedure (experienced anxiety).
  The child's anxiety level was assessed using the Visual Analog Scale for Anxiety (VAS-A), a 10 cm horizontal line scored from 0 ("no anxiety") to 10 ("worst possible anxiety"), with each point represented by a corresponding facial expression. Parents were asked to rate the child's anxiety level on the scale.

SECONDARY OUTCOMES:
Satisfaction Level | Satisfaction was measured once - immediately after the procedure.
  Both the child and the parent rated their satisfaction with the Storytelling Caterpillar on a scale from 1 ("not satisfied at all") to 10 ("very satisfied").

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Başakşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains identifiable health information of pediatric participants, and sharing is restricted to protect patient privacy in accordance with ethical and legal requirements.